CLINICAL TRIAL: NCT02995070
Title: The Influence Low Intensity Laser Therapy (LILT) in Connective Tissue Graft for Root Coverage in Smokers. A Controlled Clinical Trial
Brief Title: Low Intensity Laser Therapy in Connective Tissue Graft for Root Coverage in Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF 7
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTG + LLLT (Experimental): The irradiation will be performed with a GaAlAs diode laser that will continuously emits a wavelength of 660 nm with a power of 30 milliwatts. The patients allocated for the LLLT group will receive the following protocol for laser application: Five (5) points of irradiation will be performed using a total energy density (fluence) of 15 J/cm2 and a time of 20 seconds. During irradiation, the tip of the laser probe will be placed perpendicularly with slight contact on the area. Laser therapy will be initiated in the immediate postoperative period (just after sutures) and will be repeated by seven more applications performed every other day, with a total of 8 laser applications. The power of the equipment will be calibrated prior to each application.
  Interventions: Procedure: CTG; Device: LLLT
- CTG + SHAM (Sham Comparator): The patients allocated to the control group will receive sham irradiation. For this, black rubber protection will be placed at the tip of the laser device, which will not allow the light to reach the tissue. The applications will be performed by a different operator from the one who will measure the study parameters. During irradiation, the tip of the laser probe will be placed perpendicularly with slight contact on the area. Laser therapy will be initiated in the immediate postoperative period (just after sutures) and will be repeated by seven more applications performed every other day, with a total of 8 laser applications.
  Interventions: Procedure: CTG; Device: SHAM

INTERVENTIONS:
Procedure: CTG — Periodontal plastic surgery for root coverage by the trapezoidal flap plus connective tissue graft
  Other Names: Periodontal plastic surgery
Device: LLLT — Low Level Laser Therapy on the buccal recipient site of connective tissue graft.
  Other Names: Low level GaAlAs laser
  Arms: CTG + LLLT
Device: SHAM — Simulation of GaAlAs laser to irradiation on connective tissue graft recipient site.
  Other Names: Low level GaAlAs laser sham
  Arms: CTG + SHAM

SUMMARY:
The aim of this study is to evaluate the influence of therapy with low-intensity laser technique associated with connective tissue graft for root coverage in smokers and compare the results with non- smokers

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Science and Technology Institute - São José dos Campos, College of Dentistry.

The selected smokers patients will be randomly allocated by a computer generated list into:

Group CTG (n=15): patients who will receive only the connective tissue graft procedure to treat gingival recession and a simulation of laser therapy application (SHAM).

Group CTG+ LLLT (n=15): patients who will receive the connective tissue graft procedure to treat gingival recession plus 8 applications of low-level-laser therapy (LLLT) to treat gingival recession.

All surgeries will be performed by the same expert periodontist. Before the surgical procedure, all patients were enlightened about the causes and consequences of gingival recession and prevention techniques. Factors related to the origin of gingival recession, such as toothbrush trauma and inflammation caused by biofilm, will be controlled through instruction on standardized brushing technique to avoid the influence of other hygiene methods capable of promoting trauma on soft tissues. Standardized dental floss and toothbrushes were given to patients. The surgical technique adopted in the recession defects was the trapezoidal-type of coronally advanced flap (CAF) and the connective tissue graft (CTG) will be removed from palate mucosa . Briefly, a first incision on the palate will be performed perpendicularly to the long axis of the teeth, 2 to 3 mm apical to the gingival margin. The mesial-distal length of the incision will be determined by the length of the graft required to cover the recession. Because the selected recessions were in maxillary canines and premolars, the lengths of the graft varied minimally (10-12mm). The second incision will be made parallel to the first one (1-2 mm apically and parallel to the long axis of the teeth) to separate the subepithelium connective tissue from the epithelial layer. The incision is carried far enough apically to provide a 7- mm height of connective tissue to cover the denuded root surface. Afterward, another incision parallel to the long axis of the teeth starting from the first incision will be performed to separate the subepithelium connective tissue from the periosteum. Then, the connective tissue graft will be removed from the palate as atraumatically as possible. Single sutures will be made on the palate (4-0 silk) and the graft will be sutured on the receptor site. The irradiation will be performed with a Gallium aluminum arsenide laser (GaAlAs) that continuously emitted a wavelength of 660 nm. Thirty milliwatts will be used for 20 seconds and the total applied energy (fluence) will be 15 Joules per cm2 (3 Joules/ per point and an application time of 4 seconds per point).

Clinical, esthetics, and comfort of patients parameters were assessed at baseline, 3 and 6 months after the procedure.

Quantitative data were recorded as mean ± standard deviation (SD), and normality was tested using Shapiro-Wilk tests. The probing depth (PD), relative gingival recession (RGR), clinical attachment level (CAL), keratinized tissue thickness (KTT), keratinized tissue width (KTW), and dentin hypersensitivity (DH) values were examined by two-way repeated measures ANOVA to evaluate the differences within and between groups, followed by a Tukey test for multiple comparisons when the Shapiro-Wilk p value was ≥ 0.05. Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using visual analog scale (VAS) were analyzed by T-tests. The frequency of complete root coverage was compared using χ2 tests. Intergroup root coverage esthetic score (RES) comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Miller class I or II gingival recession in the maxillary canines or premolars
* Visible cemento-enamel junction (CEJ) with pulp vitality;
* Patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤20%;
* Patients older than 18 years old; probing depth ˂3 mm in the included teeth;
* Patients who agreed to participate and signed an informed consent form.

Exclusion Criteria:

* Patients presenting systemic problems that would contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers or pregnant women;
* Patients who underwent periodontal surgery in the area of interest;
* Patients with orthodontic therapy in progress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of defect coverage | 6 months

SECONDARY OUTCOMES:
Root coverage esthetic score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- Felipe Lucas da Silva Neves, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia VG, Macarini VC, de Almeida JM, Bosco AF, Nagata MJ, Okamoto T, Longo M, Theodoro LH. Influence of low-level laser therapy on wound healing in nicotine-treated animals. Lasers Med Sci. 2012 Mar;27(2):437-43. doi: 10.1007/s10103-011-0956-4. Epub 2011 Jul 13. PMID 21750957
- [Background] Ozturan S, Durukan SA, Ozcelik O, Seydaoglu G, Haytac MC. Coronally advanced flap adjunct with low intensity laser therapy: a randomized controlled clinical pilot study. J Clin Periodontol. 2011 Nov;38(11):1055-62. doi: 10.1111/j.1600-051X.2011.01774.x. Epub 2011 Sep 15. PMID 22092477
- [Background] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056